CLINICAL TRIAL: NCT05165043
Title: Position Changes in Endoscopic Cirrhosis Variceal Hemorrhagic Spot Detection: a Retrospective Study of 11 Cases
Brief Title: Position Changes in Cirrhosis Hemorrhagic Spot Detection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PC-1.0
Record Dates: First submitted 2021-11-29; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Emergency Hemostasis
Keywords: Complications of cirrhosis; Variceal bleeding; Position change; Emergency hemostasis; Rebleeding

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PC group: The patients who conducted position change due to massive EGVB resulting in poor visualization in the stomach were included. The patients were characterized in terms of age, sex, causes of liver cirrhosis, adverse events (AEs) during position change, additional findings after body position change, treatment regimens and follow-up information.
  During position changing procedure, endoscopist withdrew the gastroscope from the stomach and patients changed from the left lateral position to the right lateral position with the help of the nurses. Then endoscopist reinserted the gastroscope into the stomach and tried to detect the addition varices after position change.
  Bleeding varices were treated by injection of N-butyl-Cyanoacrylate glue (glub B or Beltran, Compex) or/and Lauromacrogol (Shanxi, Tianyu).
  Interventions: Procedure: position change

INTERVENTIONS:
Procedure: position change — The patients who conducted position change due to massive EGVB resulting in poor visualization in the stomach were included,patients changed from the left lateral position to the right lateral position.

SUMMARY:
The patients who conducted position change due to massive EGVB resulting in poor visualization in the stomach were included. Those with incomplete information were excluded. The patients were characterized in terms of age, sex, causes of liver cirrhosis, adverse events (AEs) during position change, additional findings after body position change, treatment regimens and follow-up information.

DETAILED DESCRIPTION:
The patients who conducted position change due to massive EGVB resulting in poor visualization in the stomach were included. Those with incomplete information were excluded. The patients were characterized in terms of age, sex, causes of liver cirrhosis, adverse events (AEs) during position change, additional findings after body position change, treatment regimens and follow-up information.

The gastroscopes procedure was started in the left lateral position in all patients. Bleeding varices detected before the position change were stopped by the endoscopic hemostatic measures described above. The following conditions would consider a change of position during gastroscopy: (1) A large amount of blood or blood clot was found after reaching the stomach, making it difficult to suction adequately which led to poor mucosal visuality; (2) Persistent massive bleeding from a blood vessel that filled the stomach cavity rapidly after suction, making it impossible to clarify the bleeding vessel.During position changing procedure, endoscopist withdrew the gastroscope from the stomach and patients changed from the left lateral position to the right lateral position with the help of the nurses. Then endoscopist reinserted the gastroscope into the stomach and tried to detect the addition varices after position change.

Bleeding varices were treated by injection of N-butyl-Cyanoacrylate glue (glub B or Beltran, Compex) or/and Lauromacrogol (Shanxi, Tianyu).

ELIGIBILITY:
Inclusion Criteria:

* conducted position change due to massive EGVB resulting in poor visualization in the stomach

Exclusion Criteria:

* incomplete information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who conducted position change due to massive EGVB resulting in poor visualization in the stomach were included.
Sampling Method: Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2021-12-30 (Estimated); Primary Completion 2022-01-05 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of successful hemostasis | within 5 days
  non-rebleeding within 5 days after treatment
Incidence of rebleeding | within 5 days
  early rebleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo first hospital, Ningbo, Zhejiang, China